CLINICAL TRIAL: NCT02291406
Title: Importance of Surgical Approach for Hysterectomies on Metabolic Effects Regarding Development of Insulin Resistance and Subsequent Recovery. A Randomized Controlled Study.
Brief Title: Importance of Surgical Approach for Gynecological Surgery on Metabolic Effects and Subsequent Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Kerstin Nilsson MD, PhD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLL-431061
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-10

CONDITIONS: Insulin Resistance
Keywords: Hysterectomy; Insulin resistance; Metabolism
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot assisted laparoscopic hysterectomy (Active Comparator): Robot assisted laparoscopic total hysterectomy
  Interventions: Procedure: Robot assisted laparoscopic hysterectomy
- Abdominal hysterectomy (Active Comparator): Standard extrafascial abdominal total hysterectomy through a low transverse abdominal wall incision.
  Interventions: Procedure: Abdominal hysterectomy

INTERVENTIONS:
Procedure: Abdominal hysterectomy — Standard extrafascial abdominal total hysterectomy through a low transverse abdominal wall incision.
  Arms: Abdominal hysterectomy
Procedure: Robot assisted laparoscopic hysterectomy — Robotic assisted total laparoscopic hysterectomy.
  Arms: Robot assisted laparoscopic hysterectomy

SUMMARY:
Insulin resistance is a key reaction to surgery and trauma and reflects the degree of metabolic stress. With greater degree of insulin resistance the development of complications increase, in particular infectious complications. The aim of this study is to determine if robotic assisted total laparoscopic hysterectomy induces less insulin resistance compared to abdominal hysterectomy. Insulin resistance is measured by the hyperinsulinemic normoglycemic clamp method. In addition inflammatory factors and clinical recovery will be measured.

DETAILED DESCRIPTION:
This is a prospective randomized controlled single center study. Primary screening will take place in the gynecological ward of Orebro University hospital according to the inclusion and exclusion criteria. 20 patients will be enrolled. All participants are randomized between robotic assisted total laparoscopic hysterectomy and total abdominal hysterectomy.

The main purpose of this study are to determine if robotic assisted laparoscopic hysterectomy induces less insulin resistance compare to abdominal hysterectomy. Both patients with benign and malignant disease are included. In addition inflammatory factors such as IL-6 and CRP are measured and clinical recovery is measured.

Each patient will be studied twice using the hyperinsulinemic normoglycemic clamp, a method that now is the gold standard for determining insulin sensitivity. During the clamp insulin is infused intravenously to attain an elevation at levels seen after an abnormal meal. At the same time glucose is infused to balance the effect of insulin and to maintain normal blood glucose level. The amount of the glucose infusion needed is the level of insulin sensitivity. The clamp procedure is performed before surgery as a control measure and the morning after surgery to yield the relative change in insulin sensitivity caused by the operation (postoperative insulin resistance). Before the onset of the infusion, and after 60 minutes of steady state during insulin stimulation, blood is collected for the analysis of immune function. This is also collected 3 hours after surgery.

A 6 minutes walk test is performed before surgery and the day after surgery, in order to determine a more clinical measure on recovery.

In addition demographic and clinical data are systematically collected during the hospital stay and 30 days after.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Scheduled to total hysterectomy and/or bilateral salpingo-oophorectomy (BSOE).
* Both malignant or benign indications
* The operation should be technically possible to perform with laparoscopy or by abdominal incision, including approval from an anesthesiologist
* Acceptance to participate in the study and signed written informed consent document
* Proficiency in Swedish language

Exclusion Criteria:

* The operation is anticipated to comprise more than the hysterectomy + BSOE
* Diabetes mellitus
* Severe chronic pain or massive pain medication
* Severe inflammatory disease like active severe endometriosis or inflammatory bowel disease
* Known severe adhesions in the abdomen
* Contraindications on non steroidal analgesia
* Medication with drugs or disease affecting insulin resistance for example cortisone
* Mentally disabled women who cannot fill in the questionnaires or understand the consequences of participating in a trial
* Severe psychiatric disease or on medication for psychiatric disease so that the physician consider participation in the trial inappropriate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | 3 weeks
  Insulin resistance is measured by the hyperinsulinemic normoglycemic clamp, a method that now is the golden standard for determining insulin sensitivity. The clamp is measured 1-2 weeks before surgery and on the morning after surgery.

SECONDARY OUTCOMES:
Changes in biomarkers of inflammation and the immune system. | 3 weeks
  Biomarkers for example IL6 and CRP are measured. Biomarkers are measured two times during the hyperinsulinemic normoglycemic clamp before surgery, 3 hours after surgery and two times during the clamp after surgery.
6 minutes walk test | 3 weeks
  Measured before surgery and on the day after surgery 25-26 hours after surgery.
postoperative outcomes | 4 weeks
  Postoperative outcome is registered systematically according to the ERAS Society register.
complications | 4 weeks
  Adverse events are registered systematically from start of anesthesia to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Nilsson, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, Örebro University Hospital, School of medicine, Örebro University, Sweden; Lena Wijk, MD, Principal Investigator — Department of Obstetrics and Gynecology, Örebro University Hospital, School of Health and Medical Sciences, Örebro University, Sweden; Olle Ljungqvist, MD, Prof, Study Chair — Department of Surgery, Örebro University Hospital, School of Health and Medical Sciences Örebro University, Sweden.
Locations (1):
- Örebro Univeristy Hospital, Örebro, Sweden

REFERENCES:
- [Derived] Wijk L, Nilsson K, Ljungqvist O. Metabolic and inflammatory responses and subsequent recovery in robotic versus abdominal hysterectomy: A randomised controlled study. Clin Nutr. 2018 Feb;37(1):99-106. doi: 10.1016/j.clnu.2016.12.015. Epub 2016 Dec 23. PMID 28043722